CLINICAL TRIAL: NCT05618431
Title: Prospective Biological Sample Collection Aiming to Validate Non-invasive Prenatal Tests by Analyzing Fetal DNA Present in Maternal Blood Using a Next-generation Digital PCR Technique
Brief Title: Validate Non-invasive Prenatal Tests for the Detection of Chromosomal Abnormalities
Acronym: NIPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A00290-43
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Validation of New Test NIPT
MeSH Terms: interventions — dichlorobis(azomycin)platinum II

STUDY DESIGN:
Intervention Model Description: Demonstrating non-inferiority means ensuring that the product tested does not have an efficacy that would be too inferior to the reference product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pregnant women (Other): Pregnant woman 18 and 50 years oldbetween 10 and 40 weeks of pregnancy
  Interventions: Other: NIPT

INTERVENTIONS:
Other: NIPT — This research aims to develop and validate a new method for non-invasive prenatal testing

SUMMARY:
This study will be conducted on pregnant patients for whom there is a suspicion of a chromosomal abnormality of the fetus. These are patients eligible for non-invasive prenatal screening as part of their usual pregnancy surveillance. This research aims to develop and validate a new method for non-invasive prenatal testing.

This prospective collection study will allow the collection of biological samples necessary for the development, testing and validation of these new tests

DETAILED DESCRIPTION:
The main objective : of the study is the validation of non-invasive prenatal tests for the detection of chromosomal abnormalities by analyzing the fetal DNA present in maternal blood by a new generation digital PCR.

The secondary objective of this research: is to validate the reliability of the test on both populations (affected and unaffected) and its ability to detect the following anomalies: Triple X and 22q.11.2 Micro-deletion.

Type and methodology of research :

Although the only act of the research being the sampling of a maximum of 3 additional blood tubes for a maximum volume of 30 mL during a blood test as part of the care, this study is qualified as research involving the human person at risk and minimal constraints.

Provisional research calendar :

The inclusion period for subjects is 18 months, from the date of inclusion of the first patient.

The duration of the subjects' participation in this research protocol is related to the time of inclusion and the procedure of blood collection by venipuncture.

The end of participation of patients included in the study is effective as soon as the collection of the sample is completed.

Primary endpoint:

Evaluation of the non-inferiority of a new non-invasive test for the detection of chromosomal abnormalities and to determine the accuracy of fetal sex classification by the new NIPT method combined with next-generation digital PCR from acellular fetal DNA found in maternal plasma.

Secondary endpoint:

Evaluation of test performance in both populations (affected and unaffected) Evaluation of the performance of the test to detect the following anomalies: Triple X and 22q.11.2 Micro-deletion.

ELIGIBILITY:
Inclusion criteria

1. Pregnant woman between 10 and 40 weeks of pregnancy 2. Gestational age at time of collection of the known sample 3. Maternal age 18-50 years 4. Sex of the fetus or newborn known (confirmed by doctor or karyotype) 5. Number of known fetuses 6.a) for affected samples: result of the karyotype available 6.b) for unaffected samples: preferably, result of the available karyotype; A secondarily negative NIPT result associated with a doctor's confirmation of the delivery of a healthy baby.

7. Have a diagnostic result (such as amniocentesis or CVS) available if NIPT is positive 8. Patients Affiliated to a social security scheme or entitled to.

Non-inclusion criteria

1. Confirmed mosaic sample
2. Confirmed maternal mosaicism
3. Recent maternal blood transfusion known
4. Patient who received an organ transplant
5. Patient who underwent surgery
6. Patient on immunotherapy or stem cell therapy and/or other maternal malignancy
7. Patient already included in the study during pregnancy
8. Patient under guardianship or curatorship or safeguard of justice

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1790 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the non-inferiority of a new non-invasive test for the detection of chromosomal abnormalities by analyzing the fetal DNA present in maternal blood by a new generation digital PCR | 18 months
  As part of this study, comparative analyses will be carried out:
  For qualitative variables: Pearson's Chi ² test will be used unless the estimated theoretical number in a cell is less than five, in which case the Yates continuity correction or the exact Fisher test will be applied.
  For quantitative variables: the t-test or an analysis of Student's variance will be performed. Otherwise, post-hoc analyses will be performed using the Student-Neuman-Keuls test. If the data is not distributed normally, nonparametric tests will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided